CLINICAL TRIAL: NCT01804738
Title: Investigating Inter-individual Variability in Glycemic and Insulin Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Human Development and Potential (IHDP), Singapore (Other)
Responsible Party: Principal Investigator, Lee Yung Seng, Associate Professor, Institute for Human Development and Potential (IHDP), Singapore
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2012/01149
Record Dates: First submitted 2013-03-04; First posted 2013-03-05 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Hyperglycemia; Insulin Sensitivity
Keywords: Ethnic differences; Inter-individual variability; Glycemic response; Insulin response; Mastication; Salivary alpha-amylase; Gastric emptying; Metagenome
MeSH Terms: conditions — Hyperglycemia; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Glucose (No Intervention): Glucose anhydrous 50g dissolved in 250ml water
- Jasmine rice (Active Comparator): 50g available carbohydrate portion
  Interventions: Other: Jasmine rice
- Parboiled basmati rice (Active Comparator): 50g available carbohydrate portion
  Interventions: Other: Parboiled basmati rice

INTERVENTIONS:
Other: Jasmine rice — Standardised rice:cooking liquid ratio for 50g available carbohydrate portion
  Arms: Jasmine rice
Other: Parboiled basmati rice — Standardised rice:cooking liquid for 50g available carbohydrate portion
  Other Names: Dreamrice
  Arms: Parboiled basmati rice

SUMMARY:
This study aims to test the following hypothesis in healthy lean young men:

* There are differences in glycemic response (GR) and insulin response (IR) between Chinese, Malay and Asian-Indian
* There are differences in GI values to the same food between ethnic groups
* There are ethnic differences postprandial GR and IR for high vs low GI foods
* Mastication, salivary amylase activity, gastric emptying rate and gut microbiota composition influences inter-individual glycemic and insulinemic variability
* Ethnic differences in mastication, salivary amylase activity, gastric emptying rate and gut microbiota composition determines the inter-ethnic glycemic and insulinemic variability

DETAILED DESCRIPTION:
There is extensive evidence that numerous biological digestive factors varies between individuals and influence postprandial glycemic response (GR) and insulin response (IR), which are well established risk factors that precipitate the development of Type 2 diabetes mellitus (T2DM). However, no study to date has measured and compared physiological parameters such as mastication, salivary amylase activity, gastric emptying rates and gut microbiota in a multi-ethnic Asian population, with varying prevalence of obesity and T2DM. The aim of this study is to investigate ethnic differences in GR and IR as well as the GI values of foods. Additionally, we aim to examine how physiological digestive factors contribute to inter-ethnic and inter-individual variability in GR and IR. The study outcomes can potentially explain, in part, the varying susceptibility to obesity, T2DM and DM control between Chinese, Malays and Asian-Indians in Singapore, as reflected by the differences in prevalence of obesity, T2DM and DM control among the three local ethnic groups.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to comply with study procedures and given written informed consent
* Chinese/Malay/Indian males, aged 21-40 years old
* Body mass index (BMI) between 18.5 - 24.9 kg/m2
* Fasting blood glucose between 4 - 6 mmol/L
* Sedentary adults, with <1 episode of exercise per week
* Not have a history of food allergies or food intolerances
* Be a non-smoker
* Drinks less than 3 units of alcohol per day
* Not taking antibiotics for the past 3 weeks

Exclusion Criteria:

* Subjects with known chronic diseases, including diabetes, untreated hypertension, renal impairment, gastrointestinal problems, and other significant medical conditions
* BMI <18.5 kg/m2 or >25 kg/m2
* Fasting blood glucose ≥7.0mmol/l
* Alcohol consumption >3 drinks / day
* Use of medications known to affect glucose metabolism
* Recent changes in weight of >5% over the past 3 months
* Significant changes in diet over the past 3 months
* History of eating disorders or irregular eating habits
* Taking antibiotics medications over the past 3 weeks

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Postprandial glycemic and insulin responses | Every 15 mins in the first hour and every 30 mins for the next 2 hours after food consumption
  Capillary bloods will be obtained using finger-pricks

SECONDARY OUTCOMES:
Physiological digestive functions | Up to 5 hours
  They include: measurement of mastication rate, salivary amylase activity, gastric emptying rate and gut microbiota composition

OTHER OUTCOMES:
Glycemic index values | 180 mins
  Derivation of the glycemic index values of foods using postprandial glycemic response to reference food and test foods.

CONTACTS AND LOCATIONS:
Overall Officials: Yung S Lee, A/Prof, Principal Investigator — Institute for Human Development and Potential (IHDP), Singapore
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

REFERENCES:
- [Result] Tan VM, Ooi DS, Kapur J, Wu T, Chan YH, Henry CJ, Lee YS. The role of digestive factors in determining glycemic response in a multiethnic Asian population. Eur J Nutr. 2016 Jun;55(4):1573-81. doi: 10.1007/s00394-015-0976-0. Epub 2015 Jul 10. PMID 26160548
- [Result] Tan VM, Wu T, Henry CJ, Lee YS. Glycaemic and insulin responses, glycaemic index and insulinaemic index values of rice between three Asian ethnic groups. Br J Nutr. 2015 Apr 28;113(8):1228-36. doi: 10.1017/S0007114515000586. Epub 2015 Mar 19. PMID 25789978
- [Result] Ooi DS, Tan VM, Ong SG, Chan YH, Heng CK, Lee YS. Differences in AMY1 Gene Copy Numbers Derived from Blood, Buccal Cells and Saliva Using Quantitative and Droplet Digital PCR Methods: Flagging the Pitfall. PLoS One. 2017 Jan 26;12(1):e0170767. doi: 10.1371/journal.pone.0170767. eCollection 2017. PMID 28125683